CLINICAL TRIAL: NCT06961461
Title: AI-assisted Quality Control Study of Multimodal Data in the Epidemiological Survey of Shanghai Nicheng Cohort Study
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Huating, Professor, Shanghai 6th People's Hospital
Other Study IDs: 2025-04
Record Dates: First submitted 2025-04-29; First posted 2025-05-08 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-04

CONDITIONS: Quality Control; Cohort Studies

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Manual quality control: The questionnaire content was checked by manually listening back to the recordings and errors were recorded manually
- Use AI tools to conduct quality control: Quality control personnel use an integrated AI-assisted system to perform quality control on epidemiological survey data. The AI system automatically transcribes audio and analyzes data quality,. Quality control personnel conduct reviews based on AI prompts.
  Interventions: Other: AI-assisted quality control tool

INTERVENTIONS:
Other: AI-assisted quality control tool — In this study, quality control personnel will be randomly divided into an experimental group and a control group, and will use artificial intelligence-assisted quality control and manual quality control to conduct quality control on the data collected from the epidemiological survey.
  Experimental group: Quality control personnel will use the AI system to perform quality control on the questionnaire recordings.
  Control group: The questionnaire content was checked by manually listening back to the recordings and errors were recorded manually.
  Groups: Use AI tools to conduct quality control

SUMMARY:
This study is based on the Nicheng Cohort study. This study intends to analyze whether AI assistance can effectively improve the efficiency and accuracy of quality control of data collected in large-scale epidemiological surveys based on traditional quality control processes.

DETAILED DESCRIPTION:
This study randomly divided quality control personnel into an experimental group and a control group. The experimental group adopts AI assisted quality control: the AI system automatically transcribes the recorded text of the questionnaire, extracts keywords, analyzes the consistency of the Q&A logic, and generates quality control prompts. The quality control personnel will verify the question fragments according to the prompts and determine the qualification of the questionnaire; The control group relies entirely on manual quality control: the quality control personnel listen to the recording word by word, manually record the content, independently identify keyword omissions, logical contradictions, or terminology deviations, and ultimately determine whether the questionnaire is qualified. The core difference lies in the fact that the experimental group uses AI technology to accurately locate risk issues, reducing the burden of manual comprehensive screening, while the control group requires full manual review without targeted support.

ELIGIBILITY:
Inclusion Criteria:

1. Be proficient in using computers;
2. The person responsible for questionnaire quality control needs to have good dialect recognition ability;
3. Have a basic understanding or high acceptance of AI-assisted tools, and be able to adapt to the learning and application of new technologies
4. Be able to participate in the research throughout the process, abide by the research process, receive training, and be willing to complete quality control tasks as required.

Exclusion Criteria:

1. The person responsible for questionnaire quality control cannot understand or recognize Shanghai Nanhui dialect proficiently;
2. Unfamiliar with AI-assisted tools and difficult to accept technical operations;
3. Unable to participate in the research, receive training or complete the specified tasks due to other work or academic reasons;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Questionnaires in the Nicheng cohort
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-06-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Accuracy | From enrollment to the end of questionnaire quality control at 8 weeks
  changes in the efficiency and accuracy of quality control of data collected in large-scale epidemiological surveys with AI-assisted tool

SECONDARY OUTCOMES:
Completeness and consistency | From enrollment to the end of questionnaire quality control at 8 weeks
  AI-assisted quality control in questionnaire quality control improves the integrity and consistency of questionnaire data through automated keyword extraction and logical consistency checking.